CLINICAL TRIAL: NCT07292545
Title: Examining the Effectiveness of Video-Based Proprioceptive Home Exercise Program in Amyotrophic Lateral Sclerosis Patients
Brief Title: Video-Based Proprioceptive Exercise Program in ALS
Acronym: ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Evrim GÖZ, Assoc. Prof., Tarsus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TarsusUftr
Record Dates: First submitted 2025-07-10; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic latearl sclerosis; proprioception; video based exercise
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- video based exercise (Experimental)
  Interventions: Other: video based exercise

INTERVENTIONS:
Other: video based exercise — Description: The proprioceptive home exercises that will be presented to patients who meet the inclusion criteria and whose preliminary evaluation has been completed will be taught by a physiotherapist in a clinical setting, and all questions about the exercises will be answered. The proprioceptive home exercises program includes 60 and 120 degrees of shoulder flexion with eyes open and closed, respectively, while lying on the back, shoulder abduction, 65 and full normal joint movement limit elbow flexion with eyes open and closed, respectively, while lying on the back, hip and knee flexion with eyes open and closed, respectively, 90 degrees of knee flexion with eyes open and closed, respectively, while sitting, 45 and 90 degrees of knee flexion with eyes open and closed, respectively, forward and side reaching movements in the sitting position, and sitting position, eyes open and then eyes closed, for 1 minute. All patients will be asked to perform these exercises. For patients who c

SUMMARY:
In the project, it was aimed to evaluate the proprioceptive system in the disease, which is still mysterious and therefore has no curative treatment under current conditions, and to examine the effects of the video-based proprioceptive home exercise programme on trunk and limb control and daily life activity as well as trunk and limb control. The study was planned to include 20 patients with a definite diagnosis of ALS. Proprioceptive sensory examination will be performed again in these patients, who are currently being followed up with ALS diagnosis and whose physical examination including neurological examination has been performed in detail, and the "Revised Amyotrophic Lateral Sclerosis Functional Rating Scale" (R-ALSFRS) will be applied to the patients. Subsequently, the patients will be followed up by applying a video-based proprioceptive home exercise programme 3 days a week for 8 weeks. At the end of the 8th week, a detailed neurological examination including proprioceptive sensation will be performed and the R-ALSFRS scale will be applied. In addition, ALS quality of life scale will be applied to the patients before and after the home programme. The data obtained after the treatment programme will be analysed and interpreted.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disease characterised mainly by degeneration of upper and lower motor neurons. In recent years, the disease paradigm has changed and ALS has been increasingly recognised as a multi-systemic disease in which the sensory system is also affected rather than a disease limited to motor neurons. The proprioceptive system is the primary sensory system that is vital in managing motor control. Recent studies suggest that sensory impairment may occur early in ALS and that there is degeneration in proprioceptive sensory neurons. However, in the current literature, there is no study that clinically evaluates proprioception in ALS patients or provides proprioceptive training to patients. In addition, progressive muscle degeneration is frequently seen in the trunk and distal muscles in ALS, which negatively affects trunk control and leads to a decrease in the independence of patients in daily life activities and thus quality of life. In the project, it was aimed to evaluate the proprioceptive system in the disease, which is still mysterious and therefore has no curative treatment under current conditions, and to examine the effects of the video-based proprioceptive home exercise programme on trunk and limb control and daily life activity as well as trunk and limb control. The study was planned to include 20 patients with a definite diagnosis of ALS. Proprioceptive sensory examination will be performed again in these patients, who are currently being followed up with ALS diagnosis and whose physical examination including neurological examination has been performed in detail, and the "Revised Amyotrophic Lateral Sclerosis Functional Rating Scale" (R-ALSFRS) will be applied to the patients. Subsequently, the patients will be followed up by applying a video-based proprioceptive home exercise programme 3 days a week for 8 weeks. At the end of the 8th week, a detailed neurological examination including proprioceptive sensation will be performed and the R-ALSFRS scale will be applied. In addition, ALS quality of life scale will be applied to the patients before and after the home programme. The data obtained after the treatment programme will be analysed and interpreted. In the literature, the number of publications on proprioception in ALS patients is very limited. The successful completion of this project will shed light on the pathogenesis of the disease and will contribute to the planning of new researches at national and international level.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* ALS patients aged 18-70
* Those with a definite ALS diagnosis according to the Gold Coast criteria
* Those who can sit independently
* Those who have no cognitive problems
* Those who agree to participate in the study will be included in the study.

Exclusion Criteria:

* ALS patients with neurological, orthopedic or visual dysfunction mimicking ALS,
* Those who cannot complete active joint movements in the upper and lower extremities,
* ALS patients who do not agree to participate in the study will not be included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
muscle strength assesment | 1st week and 7th week
  The muscle strength assessment of ALS patients will be performed with Hoggan microFET2 (Hoggan Scientific, LLC, Salt Lake City UT, USA). It is a hand-held dynamometer. Patients are asked to perform the movement at maximum force without using a compensation mechanism, and the researcher applies resistance in the opposite direction of the movement without creating any movement in the joint, in a way that creates isometric contraction. The strength of the hip flexor, quadriceps femoris, shoulder flexor, elbow extensor, elbow flexor, trunk extensor and flexor muscles will be evaluated. 3 measurements will be taken for each muscle group and the average will be taken. There will be a 30-second rest period between measurements. The evaluations will be made by the physiotherapist.
proprioception assessment | 1st week and 7th week
  For proprioception assessment, upper extremity position sense, lower extremity position sense and trunk position sense will be assessed. Assessment of position sense J-Tech™ dual Inclinometer will be used to assess position sense. Participants will be asked to stand in a static position. For upper extremity position sense, measurements will be made in 3 separate tests with the shoulder at 60 degrees of flexion, 60 degrees of abduction and the elbow at 65 degrees of flexion. First, individuals will be asked to learn the target angle with their eyes open, then they will be asked to find the target angle with their eyes closed. Both extremities will be measured with an inclinometer and recorded. Each measurement will be performed 3 times and the average of the 3 measurements will be used for the final analysis. The knee joint will be evaluated for lower extremity position sense measurement. The knees of the errors will be flexed to 60 degr
functional status | 1st week and 7th week
  Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (R-ALSFRS) This scale, which determines the functional status of ALS patients, is the most frequently used scale in daily practice and in studies on the subject and consists of 12 headings, each scored between 0-4. While a functionally normal patient receives 48 points, the scores decrease downward due to functional deterioration. The Turkish validity and reliability study of the scale was conducted by Koç et al.

SECONDARY OUTCOMES:
Trunk control | 1st week and 7th week
  To evaluate trunk control, the Trunk Impairment Scale and the postural sway assessment in the sitting position will be performed. Trunk Impairment Scale: The Trunk Impairment Scale, developed by Verheyden et al., evaluates static and dynamic sitting balance and trunk coordination in the sitting position. The total score that can be obtained varies between 0 for minimum performance and 23 for good performance. Postural sway assessment: Postural sway assessment in the sitting position will be evaluated with GyKo (Microgate, Bolzano, Italy), which is used in movement analysis. The device performs acceleration measurement and transfers simplified data with scientifically validated algorithms directly to the computer via Microgate software, allowing real-time measurement. The GyKo sensor will be fixed to the person's torso with the help of attachment straps at the T1-T2 thoracic vertebrae level. After the patients sit on a stool suitable for their height, they are
QoL | 1st week and 7th week
  The Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) will be used to assess quality of life in ALS patients. It is a 40-question scale developed to assess quality of life in patients with ALS. The scale consists of 5 sub-dimensions: mobility, activities of daily living (ADL), eating and drinking, communication, and emotional functioning. The lowest score that can be obtained from the scale is 0, the highest score is 100, with a high score indicating poor quality of life .

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, TARSUS, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided